CLINICAL TRIAL: NCT04973397
Title: Vascular Events In Patients Undergoing Same-day Noncardiac Surgery (VALIANCE) Study - A Prospective Observational Cohort Study Evaluating Major Cardiovascular and Adverse Events in Patients Undergoing Elective Same-day Noncardiac Surgery
Brief Title: Vascular Events In Patients Undergoing Same-day Noncardiac Surgery (VALIANCE) Study
Acronym: VALIANCE
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Université de Montréal (Other); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Sponsor
Other Study IDs: MP-02-2022-9889
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Preoperative Care; Surgery--Complications; Myocardial Infarction
Keywords: Preoperative Care; Surgery; Postoperative complications; Same-day surgery; Ambulatory surgery; Outpatient surgery
MeSH Terms: conditions — Myocardial Infarction; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proportion of noncardiac surgeries performed as same-day surgery is increasing worldwide, with more complex surgeries being performed on higher risk patients in the outpatient setting. Little is known on the risk factors, incidence and prognosis of patients undergoing same-day noncardiac surgery. The main objective of this study is to inform on the incidence and risk factors of cardiovascular and other adverse events after same-day surgery and to develop risk prediction tools to better inform on the risk and selection of patients undergoing same-day surgery.

DETAILED DESCRIPTION:
The VALIANCE Study is a 15,000 patient, multicentre, prospective observational cohort of adults undergoing elective same-day noncardiac surgery and who will be followed for 90 days after surgery. The primary objective of the study is to determine the incidence of major cardiovascular complications after same-day surgery. Patients will also be followed for the occurence of other adverse postoperative complications and determine their change in quality of life at 90 days after surgery. VALIANCE will inform on the risk factors for postoperative complications and allow to develop risk prediction tools to guide patient selection and risk stratification of patients undergoing same-day surgery. The study will also look at validating the use of the Duke Activity Status Index questionnaire, Clinical Frailty Scale, and the Revised Cardiac Risk Index. Postoperative pain will be evaluated using the Brief pain inventory score and quality of life using the EQ-5D-5L questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 45-64 years of age with at least one risk factor, or ≥65 years of age;
* undergoing elective noncardiac same-day surgery;
* planned duration in the operating room 60 minutes or more;
* provided written consent.

Exclusion Criteria:

* intervention does not require the presence of an anesthesiologist;
* procedure is performed by a nonsurgical specialty (e.g., gastroenterology, pneumology, radio-oncology or radiology);
* intervention is an ophthalmologic procedure;
* previously enrolled in the VALIANCE study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible adults undergoing elective same-day noncardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Unplanned healthcare utilization | 90 days
  the number of patients who have at least one of the following: unplanned admission after surgery, unplanned outpatient visit, emergency room visit and rehospitalization after same-day surgery

SECONDARY OUTCOMES:
unplanned admission | 90 days
  the number of patients who have to be admitted to the hospital after undergoing a surgery planned as same-day
unplanned outpatient visit | 90 days
  the number of patient who had a medical visit in an outpatient setting after undergoing same-day surgery
emergency room visit | 90 days
  the number of patients who visited the emergency room without subsequent hospitalization after undergoing same-day surgery
re-hospitalization | 90 days
  the number of patients who have to be readmitted to the hospital after being discharged home following their same-day surgery
major cardiovascular complications | 90 days
  the number of patients who have at least one of the following: myocardial injury or infarction, non-fatal cardiac arrest, coronary revascularization, stroke, transient ischemic attack, new clinically significant arrythmia, congestive heart failure, unplanned postoperative admission for vascular reasons, emergency room visit for vascular reasons, rehospitalization for vascular reasons, and all-cause mortality
myocardial injury after noncardiac surgery (MINS) | 90 days
  the number of patients who experience a MINS
myocardial infarction | 90 days
  the number of patients who experience a myocardial infarction
non-fatal cardiac arrest | 90 days
  the number of patients who experience a non-fatal cardiac arrest
coronary revascularization | 90 days
  the number of patients who undergo coronary revascularization
stroke | 90 days
  the number of patients who experience a stroke
transient ischemic attack | 90 days
  the number of patients who experience a transient ischemic attack
new clinically important arrythmia | 90 days
  the number of patients who experience a new clinically important arrythmia
acute congestive heart failure | 90 days
  the number of patients who experience an acute congestive heart failure episode
deep vein thrombosis | 90 days
  the number of patients who experience a deep vein thrombosis
pulmonary embolism | 90 days
  the number of patients who experience a pulmonary embolism
major postoperative and life-threatening bleeding | 90 days
  the number of patients who experience a major postoperative and/or life-threatening bleeding
postoperative infection | 90 days
  the number of patients who experience a postoperative infection
acute kidney injury | 90 days
  the number of patients who experience a acute kidney injury
quality of life score on the 5-level EQ-5D version (EQ-5D-5L) questionnaire | 90 days
  score on the EQ-5D-5L questionnaire on 4 health profiles (level 1 to 5), overall self-rated health status (0-100 visual analogue scale), and EQ-5D-5L index value (0.01-0.99)
functional capacity score on the Duke Activity Status Index (DASI) | 90 days
  change in the score on the Duke Activity Status Index (DASI) questionnaire (0 to 58.2 points)
frailty | 90 days
  change in the level on the Clinical Frailty Scale (level 1 to 9)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Duceppe, MD, PhD, Principal Investigator — Centre Hospitalier de l'Universite de Montreal (CHUM)
Locations (16):
- United States (5):
  - Wake Forest Baptist Medical Centre, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation Fairview Campus, Cleveland, Ohio
  - Cleveland Clinic Foundation Main Campus, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center UT Health, Houston, Texas
- Canada (9):
  - St-Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - St-Micheal's Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- Maasstad Ziekenhuis Rotterdam, Rotterdam, Netherlands
- Hospital Clinic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boko MF, Khanna AK, D'Aragon F, Spence J, Conen D, Patel A, Ayad S, Wijeysundera DN, Choiniere M, Sessler DI, Carrier FM, Harlock J, Koopman JSHA, Durand M, Bhojani N, Turan A, Page G, Devereaux PJ, Duceppe E; VALIANCE Study Collaborators. Incidence and Risk Factors of Chronic Postoperative Pain in Same-day Surgery: A Prospective Cohort Study. Anesthesiology. 2024 Aug 1;141(2):286-299. doi: 10.1097/ALN.0000000000005030. PMID 38669010